CLINICAL TRIAL: NCT04715321
Title: Computed Tomography Perfusion Parameters Predict Vascular Pattern in Hepatocellular Carcinoma: A Prospective Study
Brief Title: CT Perfusion Parameters Predict Vascular Pattern in Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Other Study IDs: SCT-01
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; CT perfusion parameters; vascular pattern
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: HCC patients enrolled in our study underwent a perfusion CT examination before surgery . We used CT perfusion parameters to predict the vascular pattern of tumors.
  Interventions: Other: CT perfusion examination
- Validation cohort: HCC patients who would undergo a perfusion CT examination before surgery will be enrolled in our study from January 15, 2021. We use CT perfusion parameters to predict the vascular pattern of tumors.
  Interventions: Other: CT perfusion examination

INTERVENTIONS:
Other: CT perfusion examination — CT perfusion was performed with a 64-section multidetector CT scanner. The following CT parameters were used to acquire dynamic data: blood flow (BF), blood volume (BV), mean transit time (MTT), permeability-surface area product (PS), hepatic artery ejection fraction (HAF), hepatic artery perfusion (HAP), and hepatic portal vein perfusion (PVP). And we used these parameters to predict the vascular pattern.

SUMMARY:
Distinct vascular patterns (ECTC or Non-ECTC) of tumors plays an important role in tumor migration, metastasis and drug resistant in hepatocellular carcinoma (HCC). However, there is no non-invasive method to predict vascular pattern in clinical. In the present study, we prospectively assess CT perfusion parameters for evaluation of the vascular pattern in HCC.

ELIGIBILITY:
Inclusion Criteria:

1. age over than 18 years old
2. tumor size of less than 5 cm
3. Child-Pugh A class liver function
4. an Eastern Cooperative Oncology Group performance status of 0
5. no previous treatment for HCC
6. pathological diagnosis of hepatocellular carcinoma
7. adequate organ function (white blood cell count ≥3.0 × 109/L, absolute neutrophil count ≥1.5 × 109/L, platelet count ≥75 × 109/L, aspartate transaminase and alanine transaminase≤5 × upper limit of the normal, creatinine clearance rate of ≤1.5 × upper limit of the normal, and left ventricular ejection ≥45%)

Exclusion Criteria:

1. Patients who received antitumor therapy before recurrence, including radiotherapy, transarterial chemoembolization, tyrosine kinase inhibitor, and immune checkpoint inhibitor
2. a known medical history of HIV infection
3. pregnancy or breastfeeding
4. portal vein tumor thrombosis or hepatic vein thrombosis detected by any routine imaging modality, including ultrasonography, dynamic contrast CT and MRI
5. any evidence of tumor metastasis or prior recurrence
6. hepatic decompensation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients with tumor size of less than 5 cm who would receive liver resection.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-02-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive performance of CT perfusion | 6 months
  The primary outcome of our study is to evaluate the sensitivity and specifity of CT perfusion in predicting vascular pattern of HCC

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  OS is the length of time from the date of randomization until death from any cause
Disease-free survival (DFS) | 6 months
  Disease-free survival is calculated from the date of surgery to tumor recurrence or death from any cause (or the date of the last follow-up if the patient was alive)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No